CLINICAL TRIAL: NCT05185505
Title: Atezolizumab and Bevacizumab Pre-Liver Transplantation for Patients With Hepatocellular Carcinoma Beyond Milan Criteria: A Feasibility Study
Brief Title: Atezolizumab and Bevacizumab Pre-Liver Transplantation for Patients With Hepatocellular Carcinoma Beyond Milan Criteria
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Maen Abdelrahim, MD, PhD, Pharm.B, Associate Professor of Medicine in Oncology, Houston Methodist Academic Institute, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00032239; ML43352 (Other Grant/Funding Number: Genentech, Inc.)
Record Dates: First submitted 2021-12-10; First posted 2022-01-11 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Hepatocellular Carcinoma; Hepatocellular Cancer
Keywords: Bevacizumab; atezolizumab; Neoadjuvant Therapy; Liver Neoplasms; Liver Transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Atezolizumab + Bevacizumab (Experimental): Patients will receive transarterial chemoembolization (TACE) every 3 months, with a maximum of 4 treatments, plus atezolizumab combined with bevacizumab.
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Atezolizumab — 1200 mg administered every three weeks for up to 6 months (up to 8 cycles) during the liver transplant waiting period
  Other Names: Tecentriq
Drug: Bevacizumab — 15 mg/kg administered every three weeks for up to 6 months (up to 8 cycles) during the liver transplant waiting period
  Other Names: Avastin

SUMMARY:
Patients with hepatocellular carcinoma (HCC) beyond Milan Criteria (MC) who are transplant-eligible will be treated with 6 months of neoadjuvant/downstaging atezolizumab plus bevacizumab while receiving standard of care transarterial chemoembolization (TACE). We hypothesize that atezolizumab and bevacizumab can appropriately bridge patients with HCC beyond MC to transplantation and not increase the risk of 1-year post-transplant rejection.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) represents the second most common cause of cancer-related death and accounts for over 80% of primary liver cancers worldwide.(1) Curative treatment options include surgical resection in patients with well compensated liver function and radio frequency ablation in small tumors. However, in 90% of patients, HCC occurs in the setting of cirrhosis(2) where optimal management remains liver transplantation (LT) with 5-year survival rates of approximately 80%.(3) Despite the success of LT in treating HCC, only a small portion of patients fit into standard Milan Criteria to receive a LT due to 1) advanced-stage disease and/or large tumor size preventing/delaying organ allocation and 2) a lack of neoadjuvant (bridging) therapies that can effectively down-stage or delay tumor progression for patients while on the LT waiting list. The proposed clinical trial will evaluate the feasibility of using a combination of the chemotherapeutic interventions atezolizumab(4) and bevacizumab(5) in a group of patients with HCC who have tumors beyond the Milan Criteria (in brief, 5 - 10 cm), in order to appropriately bridge them to liver transplantation without increasing the risk of graft rejection within 1-year post-LT.

Globally, Milan Criteria (MC),(6) defined as one single tumor < 5cm or 3 tumors < 3cm, is the most commonly recognized criteria for selecting patients for deceased donor LT. However, it is increasingly recognized that these criteria may be restrictive and not always reflect biology of the disease.(3) Variable extended strategies have been employed including the i) extended Toronto Criteria(7) (where no limitation in tumor burden is imposed provided the tumor is not poorly differentiated and there is no evidence of extrahepatic disease or vascular invasion), ii) Ontario criteria, where patients are eligible based on Total Tumor Volume (TTV, ≤ 145cm^3) and alpha fetoprotein (AFP < 1000 ng/mL), or iii) University of California San Francisco criteria (tumor size ≤6.5 cm) and beyond.

A number of centers have implemented downstaging strategies incorporating AFP dynamics to help select who may benefit.(8) Despite similar survival in patients beyond MC successfully receiving a transplant,(7) a considerably higher rate of drop-off from the waiting list exists and survival in this population is particularly poor.(9) Downstaging patients to MC and transplant most commonly involves locoregional therapies (LRT); however, for patients who do not reach transplant, the long term survival after receiving systemic treatments is low.

The IMbrave150 study of atezolizumab and bevacizumab versus sorafenib demonstrated response rates of 29.8% vs 12%, respectively, and median overall survival of 19.8 months in the combination arm versus 13.4 months in the sorafenib alone arm (HR 0.66, 95% CI 0.52, 0.85; p=0.0009).(10) The synergistic effect of an antiangiogenic plus immune checkpoint inhibitor (CPI) can reactivate the intra-tumoral trafficking of cytotoxic T cells and create a favorable immune microenvironment for CPI antitumoral activity.(11)

This study has now shifted the treatment paradigm in HCC, suggesting a new standard of care in intermediate stage HCC refractory to local therapies and those with advanced stage disease eligible for first line treatment.(12) This data highlights the importance of systemic treatment in the management of HCC and challenges historical treatment paradigms. It further emphasizes the need to maintain liver function so that patients can receive systemic therapies.

There is little data to support systemic treatments both in the neoadjuvant setting and as a bridging or downstaging strategy to liver transplantation. Continued eligibility and timing of transplantation are crucial factors which can be influenced by donor availability, Model for End-stage Liver Disease (MELD) score and blood group. A recent case report has, however, demonstrated the feasibility of PD-1 blockade prior to orthotopic liver transplantation with no evidence of disease recurrence 1-year post-transplant. Nivolumab (OPDIVO, Bristol-Myers Squibb Co., Princeton, NJ USA)(13) was stopped in this case 6 weeks prior to transplant.(14) The half-life of 27 days for atezolizumab and 20 days for bevacizumab suggests a need to stop at a similar time point when using atezolizumab/bevacizumab.

Atezolizumab (TECENTRIQ®, Genentech, Inc., South San Francisco, CA) is a humanized immunoglobulin (Ig) G1 monoclonal antibody that targets PD L1 and inhibits the interaction between PD-L1 and its receptors, PD-1 and B7-1 (also known as CD80), both of which function as inhibitory receptors expressed on T cells. Therapeutic blockade of PD-L1 binding by atezolizumab has been shown to enhance the magnitude and quality of tumor-specific T-cell responses, resulting in improved anti tumor activity.(15,16) Atezolizumab has minimal binding to Fc receptors, thus eliminating detectable Fc effector function and associated antibody-mediated clearance of activated effector T cells.

Atezolizumab shows anti-tumor activity in both nonclinical models and cancer patients and is being investigated as a potential therapy in a wide variety of malignancies. Atezolizumab is being studied as a single agent in the advanced cancer and adjuvant therapy settings, as well as in combination with chemotherapy, targeted therapy, and cancer immunotherapy.

Atezolizumab is approved for the treatment of urothelial carcinoma, non-small cell lung cancer, small-cell lung cancer, liver and triple-negative lung cancer. Please refer to the Atezolizumab Investigator Brochure (IB) for details on nonclinical and clinical studies.

Bevacizumab (AVASTIN®, Genentech, Inc., South San Francisco, CA) is a recombinant humanized monoclonal IgG1 antibody that binds to and inhibits the biologic activity of human vascular endothelial growth factor (VEGF) in vitro and in vivo assay systems.

Bevacizumab was first granted marketing approval in the US on 26 February 2004 in combination with IV 5-fluorouracil-based chemotherapy for the first-line treatment of patients with metastatic carcinoma of the colon or rectum. Bevacizumab is approved in over 100 countries for one or more of the following indications: breast cancer, non-small cell lung cancer (NSCLC), renal cell cancer, glioblastoma multiforme, cervical cancer, epithelial ovarian cancer, primary peritoneal cancer, and fallopian-tube cancer.

Bevacizumab has been studied in a multitude of Phase I, II, and III clinical trials in more than 22,000 patients and in multiple tumor types. Approximately 1,720,000 patients have been exposed to bevacizumab as a marketed product or in clinical trials. Please refer to the bevacizumab Investigator Brochure for descriptions of all completed Phase I, II, and III trials reported to date.

The combination of atezolizumab and bevacizumab as first-line treatment for non-resectable or metastatic HCC was assessed for safety and efficacy in two studies: GO30140 and YO40245 (IMbrave150).

Study GO30140 investigated atezolizumab plus bevacizumab in combination as first-line therapy for patients with metastatic HCC.(17) It was a Phase Ib, multicenter, open-label study trial with many arms. Arm A evaluated patients who had not received prior systemic therapy. Arm F included 119 patients with locally advanced or metastatic HCC who were randomized 1:1 to atezolizumab plus bevacizumab or atezolizumab monotherapy as first-line therapy. Study results for Arm A demonstrated an objective response rate (ORR) assessment per Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1) of 37% (36%; 95% CI 26-46). For the patients who responded, 12 patients (12%) achieved a complete response (CR) and 25 patients (24%) achieved a partial response (PR). The combination of atezolizumab plus bevacizumab was generally well tolerated. Arm F demonstrated an objective response rate in 20% (95% CI 11-32), with 1 patient (2%) showing complete response and 11 (18%) with partial response.

Study YO40245, called IMbrave 150, was a phase III study including 501 randomized patients with unresectable HCC.10 Patients were randomized 2:1 to atezolizumab (1,200 mg intravenously every 3 weeks) plus bevacizumab (15 mg/kg intravenously every 3 weeks) or sorafenib (400 mg twice daily). The duration of their treatment extended until unacceptable toxicity or reduced clinical benefit per the study investigators. There was a significant improvement in overall survival response rates of 29.8% vs 12%, respectively, and median overall survival of 19.8 months in the combination arm versus 13.4 months in the sorafenib alone arm (HR 0.66, 95% CI 0.52, 0.85; p=0.0009). The median follow-up was 15.6 months. Median progression-free survival improved to 6.8 months (combination arm) compared to 4.3 months in the sorafenib group (HR 0.59; 95% CI 0.47-0.76, p< .0001). ORR was also significantly better in the combination group compared to sorafenib (27% vs 12% p<0.0001) based on RECIST v1.1. Similar increases were demonstrated using HCC mRECIST18 criteria (33% vs 13%, p<0.0001). A comparable amount of Grade 3 - 5 adverse events were seen between groups.

This trial will enroll patients with locally advanced HCC. Given the relatively poor prognosis and limited treatment options for these patients, this population is considered appropriate for trials of novel therapeutic candidates. The benefit-risk ratio for atezolizumab + bevacizumab is expected to be acceptable in this setting.

Encouraging clinical data emerging in the field of tumor immunotherapy have demonstrated that therapies focused on enhancing T-cell responses against cancer can result in a significant survival benefit in patients with advanced malignancies.(19-21) The PD-L1 pathway serves as an immune checkpoint to temporarily dampen immune responses in states of chronic antigen stimulation, such as chronic infection or cancer. PD L1 is an extracellular protein that downregulates immune responses through binding to its two receptors, PD-1 and B7-1. PD-1 is an inhibitory receptor expressed on T cells following T-cell activation, and expression is sustained in states of chronic stimulation.(22,23) B7-1 is a molecule expressed on antigen presenting cells and activated T cells. Binding of PD-L1 to PD-1 and B7-1 inhibits T-cell proliferation and activation, cytokine production, and cytolytic activity, leading to the functional inactivation or exhaustion of T cells.(24,25) Overexpression of PD-L1 on tumor cells has been reported to impede anti tumor immunity, resulting in immune evasion.(26) Therefore, interruption of the PD-L1 pathway represents an attractive strategy for restoring tumor-specific T-cell immunity.

The combination of atezolizumab with bevacizumab is expected to down-grade the tumor size and potentially allow patients to reach the smaller tumor criteria of MC for qualifying for exception points for a liver transplant. Even if the growth is halted and not reduced to MC, stable patients may be able to achieve liver transplant without exception points if a matching donor can be located that would not be suitable for another recipient. These extended criteria donor livers would be discarded yet have shown success in circumstances such as the purpose for the current trial.

Liver transplantation provides the life-saving benefit and curative therapy for liver-limited HCC. Although there has been some success with therapeutics and LRT management for HCC, liver transplantation provides the highest survival outcome (85% at 5-yrs).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years old at the time of signing Informed Consent Form
2. Measurable or evaluable disease per RECIST v1.1 or mRECIST of unresectable HCC outside of Milan criteria
3. Histologically proven HCC, without extrahepatic disease. Patients who consent to a fresh tissue biopsy, and under the discretion of the Investigators, will provide a baseline biopsy sample for diagnosis and correlative studies. Archival tumor tissue may be used to confirm HCC in patients who do not consent to a fresh tissue biopsy.
4. Prior remote LRT is allowed if new lesions or local disease recurrence are present
5. Must be eligible for liver transplantation, defined in Section 10.4
6. Eligible and suited to receive TACE procedure(s)
7. Child-Pugh score ≤A6
8. Eastern Cooperative Oncology Group (ECOG) score 0-1
9. Life expectancy of ≥ 6 months
10. Adequate hematological and end-organ function, defined by the following laboratory test results obtained within 14 days prior to study initiation:

    1. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
    2. Lymphocyte count ≥ 0.5 x 10^9/L (500/uL)
    3. Platelet count > 75 x 109/L
    4. Hemoglobin > 9 g/dL
    5. Total bilirubin < 1.5 x upper limit of normal (ULN)
    6. Aspartate transaminase (AST),alanine aminotransferase (ALT), and alkaline phosphatase (ALP) < 2.5 x ULN
    7. Serum albumin > 2.7 g/dL
    8. Serum creatinine < 1.5x ULN or calculated creatinine clearance < 50 ml/min
    9. Urine dipstick for proteinuria ≥ 2+ unless a 24-hour urine protein < 1 g of protein is demonstrated
    10. International normalized ratio (INR) ≤ 1.5 or partial thromboplastin time (PTT) ≤ 1.5 x ULN for patients not receiving anti-coagulation. The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or PTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least two weeks prior to the first study treatment.
11. No evidence of a Grade 2 or higher esophageal and/or gastric varices. Patients must have an esophagogastroduodenoscopy (EGD) within 6 months prior to initiating the study treatment. See Section 8.7.1.2.
12. No history of hemoptysis (≥ 1/2 teaspoon of bright red blood per episode) within 1 month of study enrollment
13. Negative HIV test at screening or transplant workup
14. Negative hepatitis B surface antigen (HBsAg) test at screening or transplant workup
15. Negative total hepatitis B core antibody (HBcAb) test at screening or transplant workup, or positive total HBcAb test followed by a negative hepatitis B virus (HBV) DNA test at screening or transplant workup. The HBV DNA test will be performed only for patients who have a negative HBsAg test and a positive total HBcAb test.
16. For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods, as defined below:

    1. Women must remain abstinent or use contraceptive methods with a failure rate of <1% per year during the treatment period and for 6 months after the final dose of atezolizumab/bevacizumab Females who receive a LT are required to maintain abstinence or contraception until the End of Study.
    2. A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (≥12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
    3. Examples of contraceptive methods with a failure rate of <1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices.
    4. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception.
17. For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a condom, and agreement to refrain from donating sperm, as defined below:

    1. With a female partner of childbearing potential or pregnant female partner, men must remain abstinent or use a condom during the treatment period and for 6 months after the final dose of atezolizumab/bevacizumab to avoid exposing the embryo. Men must refrain from donating sperm during this same period. Males who receive a LT are required to maintain these criteria until the End of Study.
    2. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient. Periodic abstinence (eg, calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of preventing drug exposure.
18. Stated willingness to comply with all study procedures and availability for the duration of the study
19. Women of childbearing potential must have a negative serum or urine pregnancy test result within 14 days prior to initiation of study treatment.

Exclusion Criteria:

1. Known fibrolamellar HCC, sacromatoid HCC, or mixed cholangiocarcinoma and HCC
2. Previous systemic therapy for HCC prior to study enrollment
3. Planned or prior multi-organ transplant or prior solid organ or allogeneic stem cell transplantation
4. History of Grade ≥4 venous thromboembolism
5. History or evidence upon physical or neurological examination of central nervous system (eg seizures) unrelated to cancer unless adequately treated with standard medical therapy. Anticonvulsants (stable dose) are allowed.
6. Moderate or severe ascites
7. History of hepatic encephalopathy
8. Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg)
9. History of hypertensive crisis or hypertensive encephalopathy
10. Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months prior to drug administration
11. Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina
12. History or evidence of inherited bleeding diathesis or significant coagulopathy at risk of bleeding (i.e., in the absence of therapeutic anticoagulation)
13. Surgical procedure (including open biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity) or significant traumatic injury within 28 days prior to initiation of study treatment, or anticipation of need for major surgical procedure during the Treatment Phase of the study

    • Core biopsy or other minor surgical procedure, excluding placement of a vascular access device within 7 days prior to initiation of study treatment. Placement of a vascular access device should be at least 2 days prior to initiation of study treatment.
14. History of abdominal fistula, gastrointestinal (GI) perforation, intra-abdominal abscess, grade 2 or higher untreated esophageal or gastric varices or active GI bleeding within 6 months prior to treatment
15. Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high risk for bleeding. Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrollment. Patients who have undergone an EGD within 6 months prior to initiating the study treatment do not need to repeat the procedure.
16. Serious, non-healing wound, active ulcer, or untreated bone fracture
17. Other malignancy within 5 years prior to randomization, except for localized cancer in situ, such as basal or squamous cell skin cancer
18. Current or recent (<10 days prior to initiation of study treatment) use of aspirin (>325 mg/day), or clopidogrel (>75 mg/day). Note: The use of full-dose oral or parenteral anticoagulants for therapeutic purpose is permitted as long as the INR and/or a PTT is within therapeutic limits (according to institution standards) within 14 days prior to initiation of study treatment and the patient has been on a stable dose of anticoagulants for ≥2 weeks prior to initiation of study treatment. Prophylactic use of anticoagulants is allowed. However, the use of direct oral anticoagulant therapies such as dabigatran (Pradaxa®) and rivaroxaban (Xarelto®) is not recommended due to bleeding risk.
19. Pregnancy (positive pregnancy test) or lactation, or intention of becoming pregnant during study treatment or within 6 months after the final dose of study drugs

    o Women of childbearing potential must have a negative serum or urine pregnancy test result within 28 days prior to initiation of study treatment.
20. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently)

    • Patients with indwelling catheters (e.g., PleurX®) are allowed
21. Uncontrolled or symptomatic hypercalcemia (ionized calcium > 1.5 mmol/L, calcium > 12 mg/dL or corrected serum calcium > ULN)
22. Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with the following exceptions:

    * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (eg, patients with psoriatic arthritis are excluded) are eligible for the study provided all following conditions are met:

      * Rash must cover < 10% of body surface area
      * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
      * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
23. History of idiopathic pulmonary fibrosis, organizing pneumonia (eg, bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
24. Active tuberculosis
25. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
26. Treatment with a live, attenuated vaccine (e.g., FluMist®) within 4 weeks prior to initiation of study treatment, or anticipation of need for such a vaccine during atezolizumab treatment or within 5 months after the final dose of atezolizumab
27. Current treatment with anti-viral therapy for HBV
28. Prior treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
29. Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment
30. Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during the Treatment Phase, with the following exceptions:

    * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after Principal Investigator confirmation has been obtained.
    * Patients who received mineralocorticoids (eg, fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study.
31. History of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
32. Known allergy or hypersensitivity to any component of the Atezlizumab and Bevacizumab formulation, such as a known hypersensitivity to Chinese hamster ovary cell products
33. Inability to comply with study and/or follow-up procedures
34. Active infection requiring IV antibiotics within 2 weeks prior to initiation.

    * Note: Placement of a vascular access device should be at least 2 days prior to initiation of study treatment.
    * Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
35. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
36. History of leptomeningeal disease
37. Evidence of abdominal free air that is not explained by paracentesis or recent surgical procedure
38. History of intra-abdominal inflammatory process within 6 months prior to initiation of study treatment, including but not limited to active peptic ulcer disease, diverticulitits, or colitis.
39. Chronic daily treatment with a nonsteroidal anti-inflammatory drug (NSAID). Occasional use of NSAIDs for the symptomatic relief of medical conditions such as headache or fever is allowed
40. Uncontrolled tumor-related pain

    * Patients requiring pain medication must be on a stable regimen at study entry.
    * Symptomatic lesions (eg, bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-01-30 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of Patients Receiving Liver Transplant Experiencing Acute Rejection | Within 1 year after liver transplant
  The proportion of liver transplant patients who have acute allograft rejection

SECONDARY OUTCOMES:
Proportion of participants who experience treatment-emergent adverse events | Within 90 days of study drug administration
  Number of patients who experience an FDA-defined adverse event due to the experimental treatment
Objective Response Rate | 6 months post study drug initiation
  Combined incidence of partial response and complete response of tumors to therapy per RECIST criteria
Proportion of participants who are removed from the liver transplant waiting list after initiating the atezolizumab/bevacizumab therapy | Through study completion, up to 4 years
  Number of participants who had been on the liver transplant waitlist but are removed
The proportion of participants who proceed to liver transplantation | Through study completion, up to 4 years
  Participants who receive a liver transplant
Proportion of the liver explant tissue containing necrotic tumors | Through study completion, up to 4 years
  Number of livers explanted during liver transplant that are found to contain necrotic tumors via pathology
Recurrence-free survival in patients receiving a liver transplant | Within 1 year after liver transplant
  Measure of how many patients experience hepatocellular carcinoma recurrence
Overall survival after liver transplant | Study enrollment to 1 year after liver transplant, time of liver transplant to 1 year after liver transplant
  Number of patients who are still alive after receiving a liver transplant (taking into account death of any cause)
Tumor biomarkers | At enrollment; at time of first dose of atezolizumab/bevacizumab; 3, 6, 9, 12, 15, 18, 21, 24, 30, 39 weeks after first dose; at time of liver transplant; 1, 6, and 12 months after liver transplant
  Measurement of alpha fetoprotein tumor biomarker from blood samples
Immune Cell Biomarkers | At enrollment; at time of first dose of atezolizumab/bevacizumab; 3, 6, 9, 12, 15, 18, 21, 24, 30, 39 weeks after first dose; at time of liver transplant; 1, 6, and 12 months after liver transplant
  Measurement of biomarkers in immune cells gathered via blood samples: 1) PD-L1+ in CD4+ and CD8+ cells and 2) FOXP3, CD127, and IL-8 in T regulatory cells

CONTACTS AND LOCATIONS:
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jemal A, Bray F, Center MM, Ferlay J, Ward E, Forman D. Global cancer statistics. CA Cancer J Clin. 2011 Mar-Apr;61(2):69-90. doi: 10.3322/caac.20107. Epub 2011 Feb 4. PMID 21296855
- [Background] Nordenstedt H, White DL, El-Serag HB. The changing pattern of epidemiology in hepatocellular carcinoma. Dig Liver Dis. 2010 Jul;42 Suppl 3(Suppl 3):S206-14. doi: 10.1016/S1590-8658(10)60507-5. PMID 20547305
- [Background] Sapisochin G, Bruix J. Liver transplantation for hepatocellular carcinoma: outcomes and novel surgical approaches. Nat Rev Gastroenterol Hepatol. 2017 Apr;14(4):203-217. doi: 10.1038/nrgastro.2016.193. Epub 2017 Jan 5. PMID 28053342
- [Background] Tecentriq [Package Insert]. South San Francisco, CA: Genentech, Inc.; 2020.
- [Background] Avastin [Package Insert]. South San Francisco, CA: Genentech, Inc.; 2020.
- [Background] Mazzaferro V, Regalia E, Doci R, Andreola S, Pulvirenti A, Bozzetti F, Montalto F, Ammatuna M, Morabito A, Gennari L. Liver transplantation for the treatment of small hepatocellular carcinomas in patients with cirrhosis. N Engl J Med. 1996 Mar 14;334(11):693-9. doi: 10.1056/NEJM199603143341104. PMID 8594428
- [Background] Sapisochin G, Goldaracena N, Laurence JM, Dib M, Barbas A, Ghanekar A, Cleary SP, Lilly L, Cattral MS, Marquez M, Selzner M, Renner E, Selzner N, McGilvray ID, Greig PD, Grant DR. The extended Toronto criteria for liver transplantation in patients with hepatocellular carcinoma: A prospective validation study. Hepatology. 2016 Dec;64(6):2077-2088. doi: 10.1002/hep.28643. Epub 2016 Jun 30. PMID 27178646
- [Background] O'Rourke JM, Shetty S, Shah T, Perera MTPR. Liver transplantation for hepatocellular carcinoma: pushing the boundaries. Transl Gastroenterol Hepatol. 2019 Jan 2;4:1. doi: 10.21037/tgh.2018.12.07. eCollection 2019. No abstract available. PMID 30854488
- [Background] Gorgen A, Rosales R, Sadler E, Beecroft R, Knox J, Dawson LA, Ghanekar A, Grant D, Greig PD, Sapisochin G. Patterns and Predictors of Mortality After Waitlist Dropout of Patients With Hepatocellular Carcinoma Awaiting Liver Transplantation. Transplantation. 2019 Oct;103(10):2136-2143. doi: 10.1097/TP.0000000000002616. PMID 30801510
- [Background] Finn RS, Qin S, Ikeda M, et al. Imbrave150: Updated Overall Survival (Os) Data from a Global, Randomized, Open-Label Phase Iii Study of Atezolizumab (Atezo) + Bevacizumab (Bev) Versus Sorafenib (Sor) in Patients (Pts) with Unresectable Hepatocellular Carcinoma (Hcc). Journal of Clinical Oncology. 2021;39(3_suppl):267-267.
- [Background] Opdivo [Package Insert]. Princeton, NJ: Bristol-Myers Squibb Company; 2018.
- [Background] Schwacha-Eipper B, Minciuna I, Banz V, Dufour JF. Immunotherapy as a Downstaging Therapy for Liver Transplantation. Hepatology. 2020 Oct;72(4):1488-1490. doi: 10.1002/hep.31234. No abstract available. PMID 32171041
- [Background] Rosenberg JE, Hoffman-Censits J, Powles T, van der Heijden MS, Balar AV, Necchi A, Dawson N, O'Donnell PH, Balmanoukian A, Loriot Y, Srinivas S, Retz MM, Grivas P, Joseph RW, Galsky MD, Fleming MT, Petrylak DP, Perez-Gracia JL, Burris HA, Castellano D, Canil C, Bellmunt J, Bajorin D, Nickles D, Bourgon R, Frampton GM, Cui N, Mariathasan S, Abidoye O, Fine GD, Dreicer R. Atezolizumab in patients with locally advanced and metastatic urothelial carcinoma who have progressed following treatment with platinum-based chemotherapy: a single-arm, multicentre, phase 2 trial. Lancet. 2016 May 7;387(10031):1909-20. doi: 10.1016/S0140-6736(16)00561-4. Epub 2016 Mar 4. PMID 26952546
- [Background] Fehrenbacher L, Spira A, Ballinger M, Kowanetz M, Vansteenkiste J, Mazieres J, Park K, Smith D, Artal-Cortes A, Lewanski C, Braiteh F, Waterkamp D, He P, Zou W, Chen DS, Yi J, Sandler A, Rittmeyer A; POPLAR Study Group. Atezolizumab versus docetaxel for patients with previously treated non-small-cell lung cancer (POPLAR): a multicentre, open-label, phase 2 randomised controlled trial. Lancet. 2016 Apr 30;387(10030):1837-46. doi: 10.1016/S0140-6736(16)00587-0. Epub 2016 Mar 10. PMID 26970723
- [Background] Lee MS, Ryoo BY, Hsu CH, Numata K, Stein S, Verret W, Hack SP, Spahn J, Liu B, Abdullah H, Wang Y, He AR, Lee KH; GO30140 investigators. Atezolizumab with or without bevacizumab in unresectable hepatocellular carcinoma (GO30140): an open-label, multicentre, phase 1b study. Lancet Oncol. 2020 Jun;21(6):808-820. doi: 10.1016/S1470-2045(20)30156-X. PMID 32502443
- [Background] Lencioni R, Llovet JM. Modified RECIST (mRECIST) assessment for hepatocellular carcinoma. Semin Liver Dis. 2010 Feb;30(1):52-60. doi: 10.1055/s-0030-1247132. Epub 2010 Feb 19. PMID 20175033
- [Background] Hodi FS, O'Day SJ, McDermott DF, Weber RW, Sosman JA, Haanen JB, Gonzalez R, Robert C, Schadendorf D, Hassel JC, Akerley W, van den Eertwegh AJ, Lutzky J, Lorigan P, Vaubel JM, Linette GP, Hogg D, Ottensmeier CH, Lebbe C, Peschel C, Quirt I, Clark JI, Wolchok JD, Weber JS, Tian J, Yellin MJ, Nichol GM, Hoos A, Urba WJ. Improved survival with ipilimumab in patients with metastatic melanoma. N Engl J Med. 2010 Aug 19;363(8):711-23. doi: 10.1056/NEJMoa1003466. Epub 2010 Jun 5. PMID 20525992
- [Background] Kantoff PW, Higano CS, Shore ND, Berger ER, Small EJ, Penson DF, Redfern CH, Ferrari AC, Dreicer R, Sims RB, Xu Y, Frohlich MW, Schellhammer PF; IMPACT Study Investigators. Sipuleucel-T immunotherapy for castration-resistant prostate cancer. N Engl J Med. 2010 Jul 29;363(5):411-22. doi: 10.1056/NEJMoa1001294. PMID 20818862
- [Background] Chen DS, Irving BA, Hodi FS. Molecular pathways: next-generation immunotherapy--inhibiting programmed death-ligand 1 and programmed death-1. Clin Cancer Res. 2012 Dec 15;18(24):6580-7. doi: 10.1158/1078-0432.CCR-12-1362. Epub 2012 Oct 19. PMID 23087408
- [Background] Blank C, Gajewski TF, Mackensen A. Interaction of PD-L1 on tumor cells with PD-1 on tumor-specific T cells as a mechanism of immune evasion: implications for tumor immunotherapy. Cancer Immunol Immunother. 2005 Apr;54(4):307-14. doi: 10.1007/s00262-004-0593-x. Epub 2004 Dec 15. PMID 15599732
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Butte MJ, Keir ME, Phamduy TB, Sharpe AH, Freeman GJ. Programmed death-1 ligand 1 interacts specifically with the B7-1 costimulatory molecule to inhibit T cell responses. Immunity. 2007 Jul;27(1):111-22. doi: 10.1016/j.immuni.2007.05.016. Epub 2007 Jul 12. PMID 17629517
- [Background] Yang H, Shi J, Lin D, Li X, Zhao C, Wang Q, Zhang L, Jiang T, Zhao S, Liu X, Jia Y, Zhang Y, Cai W, Zhou C. Prognostic value of PD-L1 expression in combination with CD8+ TILs density in patients with surgically resected non-small cell lung cancer. Cancer Med. 2018 Jan;7(1):32-45. doi: 10.1002/cam4.1243. Epub 2017 Nov 23. PMID 29168339
- [Background] Blank C, Mackensen A. Contribution of the PD-L1/PD-1 pathway to T-cell exhaustion: an update on implications for chronic infections and tumor evasion. Cancer Immunol Immunother. 2007 May;56(5):739-45. doi: 10.1007/s00262-006-0272-1. Epub 2006 Dec 29. PMID 17195077
- [Background] Llovet JM, Lencioni R. mRECIST for HCC: Performance and novel refinements. J Hepatol. 2020 Feb;72(2):288-306. doi: 10.1016/j.jhep.2019.09.026. PMID 31954493
- [Background] Lyman GH, Bohlke K, Khorana AA, Kuderer NM, Lee AY, Arcelus JI, Balaban EP, Clarke JM, Flowers CR, Francis CW, Gates LE, Kakkar AK, Key NS, Levine MN, Liebman HA, Tempero MA, Wong SL, Somerfield MR, Falanga A; American Society of Clinical Oncology. Venous thromboembolism prophylaxis and treatment in patients with cancer: american society of clinical oncology clinical practice guideline update 2014. J Clin Oncol. 2015 Feb 20;33(6):654-6. doi: 10.1200/JCO.2014.59.7351. Epub 2015 Jan 20. PMID 25605844
- [Background] Orsmond GI, Cohn ES. The Distinctive Features of a Feasibility Study: Objectives and Guiding Questions. OTJR (Thorofare N J). 2015 Jul;35(3):169-77. doi: 10.1177/1539449215578649. PMID 26594739
- [Background] Eisenhauer EA, Therasse P, Bogaerts J, Schwartz LH, Sargent D, Ford R, Dancey J, Arbuck S, Gwyther S, Mooney M, Rubinstein L, Shankar L, Dodd L, Kaplan R, Lacombe D, Verweij J. New response evaluation criteria in solid tumours: revised RECIST guideline (version 1.1). Eur J Cancer. 2009 Jan;45(2):228-47. doi: 10.1016/j.ejca.2008.10.026. PMID 19097774
- [Background] Ravelli A, Minoia F, Davi S, Horne A, Bovis F, Pistorio A, Arico M, Avcin T, Behrens EM, De Benedetti F, Filipovic L, Grom AA, Henter JI, Ilowite NT, Jordan MB, Khubchandani R, Kitoh T, Lehmberg K, Lovell DJ, Miettunen P, Nichols KE, Ozen S, Pachlopnik Schmid J, Ramanan AV, Russo R, Schneider R, Sterba G, Uziel Y, Wallace C, Wouters C, Wulffraat N, Demirkaya E, Brunner HI, Martini A, Ruperto N, Cron RQ; Paediatric Rheumatology International Trials Organisation; Childhood Arthritis and Rheumatology Research Alliance; Pediatric Rheumatology Collaborative Study Group; Histiocyte Society. 2016 Classification Criteria for Macrophage Activation Syndrome Complicating Systemic Juvenile Idiopathic Arthritis: A European League Against Rheumatism/American College of Rheumatology/Paediatric Rheumatology International Trials Organisation Collaborative Initiative. Arthritis Rheumatol. 2016 Mar;68(3):566-76. doi: 10.1002/art.39332. Epub 2016 Feb 9. PMID 26314788
- See also: Medical Dictionary for Regulatory Activities Maintenance and Support Services Organization. — https://www.meddra.org/
- See also: McClain KL;., O. E. Clinical Features and Diagnosis of Hemophagocytic Lymphohistiocytosis. — https://www.uptodate.com/contents/clinical-features-and-diagnosis-of-hemophagocytic-lymphohistiocytosis